CLINICAL TRIAL: NCT03804996
Title: A Phase 1 First-in-Human Study of Bispecific Antibody TG-1801 in Subjects With B-Cell Lymphoma
Brief Title: Study of TG-1801 in Subjects With B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-1801-101
Record Dates: First submitted 2019-01-12; First posted 2019-01-15 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: B-Cell Lymphoma
Keywords: relapsed or refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence | interventions — ublituximab; LFB-R603

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG-1801 (Experimental): Arm Description: TG-1801 will be administered once every 4 weeks (28-day) cycles. Subjects who experience disease progression after completing 6 months of single agent TG-1801 will be eligible for TG-1801 single-agent re-treatment at the discretion of the investigator.
  Interventions: Drug: TG-1801
- TG-1101 (Experimental): Arm Description: TG-1801 and ublituximab will be administered once every 4 weeks (28-day cycle) for up to 6 cycles followed by TG-1801 monotherapy.
  To explore the safety of TG-1801 in combination with ublituximab will be explored at doses below and up to the RP2D. TG-1801 intrapatient dose escalation will not be permitted in combination therapy.
  Interventions: Drug: TG-1801; Biological: Ublituximab

INTERVENTIONS:
Drug: TG-1801 — Intravenous infusion over 1 hour every 4 weeks
Biological: Ublituximab — "recombinant chimeric anti-CD20 monoclonal antibody, available in 25 mg/mL administered as an IV infusion once every 4 weeks"
  Other Names: TG-1101; LFB-R603
  Arms: TG-1101

SUMMARY:
Phase 1 first in human Study to Assess the Bispecific Antibody TG-1801 in Subjects with B-Cell Lymphoma

DETAILED DESCRIPTION:
This is an open-label, multi-center, accelerated titration design study. Planned enrollment includes 1 subject at low dose levels. Subjects will receive weekly infusions of TG-1801 in a 4 week-cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed B-cell lymphoma, relapsed to or refractory after at least one prior standard therapy. For subjects with aggressive lymphoma: those who are non-candidates for high-dose therapy or autologous stem cell transplant. Refractory is defined as disease progression during or within 6 months of the most recent prior therapy, while relapsed is defined as disease progression greater than 6 months after the most recent prior therapy.
2. Measurable disease defined as at least 1 measurable disease lesion ≥ 1.5 cm in at least one diameter by CT/CT-PET or magnetic resonance imaging (MRI) in an area of no prior radiation therapy, or in an area that was previously irradiated that has documented progression.
3. Be able to provide a core or excisional lymph node biopsy for biomarker analysis from an archival or newly obtained biopsy at Screening.
4. Adequate organ function defined as:

   1. Absolute neutrophil count (ANC) > 1,000/µL and platelet count > 75,000/µL. Platelet requirements cannot be met by use of recent transfusion (within 30 days of study treatment initiation [Cycle 1 Day 1]). Growth factor support (e.g. G-CSF) is not allowed within 2 weeks prior to treatment initiation.
   2. Total bilirubin ≤ 1.5 times the ULN, or direct bilirubin ≤ ULN for subjects with total bilirubin > 1.5 ULN.
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN if no liver involvement or ≤ 5 x the ULN if known liver involvement.
   4. Calculated creatinine (Cr) clearance (CL) > 30 mL/min (as calculated by the Cockcroft-Gault or MDRD formula, 24-hour urine Cr CL also acceptable).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Male or female ≥ 18 years of age.
7. Female subjects who are not of child-bearing potential, and female subjects of child-bearing potential who have a negative serum pregnancy test within 3 days prior to Cycle 1, Day 1. Female subjects of child-bearing potential, and male partners must consent to use a medically acceptable method of contraception throughout the study period and for 4 months after the last administration of ublituximab and 30 days after last administration of TG-1801. Men of reproductive potential may not participate unless they agree to use medically acceptable contraception.
8. Willingness and ability to comply with trial and follow-up procedures and provide written informed consent.

Exclusion Criteria:

1. Prior therapy with any agent blocking the CD47/SIRPα pathway or any previous CD19 targeting therapy, including but not limited to: antibodies, fragments, bispecific bodies, or chimeric antigen receptor (CAR) T-cells.
2. Subjects receiving cancer therapy (i.e. chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) or any investigational drug within 21 days of Day 1 of Cycle 1 (42 days for prior mitomycin C or a nitrosourea).

   a. Corticosteroid therapy started at least 7 days prior to Cycle 1 Day 1 (prednisone ≤ 10 mg daily or equivalent) is allowed as clinically warranted. Topical or inhaled corticosteroids are permitted.
3. Prior autologous stem cell transplant within 6 months. Prior allogeneic hematologic stem cell transplant within 1 year and excluded if there is active graft versus host disease.
4. Subjects who have not recovered (≤ Grade 1 or at baseline) from adverse events due to previous therapy, except for alopecia and Grade 2 neuropathy due to previous cancer therapy.

   Note: Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters defined above.
5. Any severe or uncontrolled illness or other conditions that could affect their participation in the study including, but not limited to:

   1. Symptomatic, or history of documented congestive heart failure (NY Heart Association functional classification III-IV).
   2. Myocardial infarction within 6 months of enrollment.
   3. Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident, transient ischemic attack, angioplasty, cardiac/vascular stenting within 6 months of enrollment, angina not well controlled by medication.
   4. Ongoing or active infection, except localized fungal infection of skin or nails.
6. Known active Hepatitis B (e.g. HBsAg reactive), Hepatitis C (e.g. HCV RNA [qualitative] is detected), cytomegalovirus (CMV DNA by PCR), or known history of HIV.
7. Malignancy within 2 years of study enrollment except for adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, superficial bladder cancer, or localized prostate cancer.
8. Known clinically active CNS involvement.
9. History of anaphylaxis or severe allergy to a monoclonal antibody; or known or suspected hypersensitivity to the excipients contained in the study drug formulation.
10. Lactating or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Identification of Recommended Dose | 18 months of therapy
  To determine the recommended Phase 2 dose (RP2D) by identifying dose limiting toxicity (DLT), maximum tolerable dose (MTD), and optimum biologic dose (OBD).
Characterize the Safety Profile of TG-1801 | 18 months of therapy
  To characterize the safety profile of TG-1801 alone and in combination with ublituximab by evaluating the adverse event profile.

SECONDARY OUTCOMES:
Pharmacokinetic data collection | 6 months of therapy
  To evaluate the pharmacokinetics (PK) of TG-1801 including Cmax.
Anticancer activity Evaluation | 6 months of therapy
  To evaluate the preliminary anticancer activity of TG-1801 by evaluating the single-agent arm by assessing the populations of lymphocytes by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - TG Therapeutics Investigational Trial Site, Heidelberg, Victoria
  - TG Therapeutics Investigational Trial Site, Melbourne, Victoria
  - TG Therapeutics Investigational Trial Site, Nedlands, Western Australia